CLINICAL TRIAL: NCT04677010
Title: Cycle Exercise in Wheelchair Users With Muscular Dystrophy or Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nanna Scharff Poulsen, MD, PhD-student, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-20075272
Record Dates: First submitted 2020-11-17; First posted 2020-12-21 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Muscular Dystrophies; Cerebral Palsy
Keywords: wheelchair; cycle exercise
MeSH Terms: conditions — Muscular Dystrophies; Cerebral Palsy | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: One group consisting of patients with either cerebral palsy or muscular dystrophy will do a 10 weeks run-in period with no exercise immediately followed by 10 weeks of exercise. They will be testet before and after the run-in period and after the exercise period.
Who Masked: Outcomes Assessor
Masking Description: Statistics will be made by an investigator blinded to what results are from before, in-between and after the two periods of rest and exercise respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Run-in period, patients with cerebral palsy or muscular dystrophy (No Intervention): 10 weeks of no exercise
- Exercise period, patients with cerebral palsy or muscular dystrophy (Active Comparator): 10 weeks of exercise
  Interventions: Other: Cycle exercise

INTERVENTIONS:
Other: Cycle exercise — 10 weeks of cycle exercise on a cycle ergometer with motor.
  Arms: Exercise period, patients with cerebral palsy or muscular dystrophy

SUMMARY:
Wheelchair bound patients often have pain in lower back and glutes, constipation and reduced quality of life - symptoms that exercise might ameliorate. However, in wheelchair bound patients with muscular dystrophies and cerebral palsy only very little research is done on exercise. We thus wish to investigate effects of cycle exercise in wheelchair bound patients with muscular dystrophy and cerebral palsy.

DETAILED DESCRIPTION:
Wheelchair bound patients with MD or CP live a sedentary life, and probably because of this, many experience pain in lower back and glutes, obstipation, reduced quality of life, reduced activity of daily living and social withdrawal. Exercise is likely to reduce these symptoms. However, research in exercising patients confined to a wheelchair lacks 3 things: 1) Most research is done in patients that are wheelchair bound due to stroke, and these results are not necessarily transferable to patients with MD or CP. Patients with stroke differ from patients with MD and CP since they can potentially gain walking ability again, they have had walking ability up to the stroke, they are only hemiparetic and thus have normal function in the rest of the body, their muscles are atrophic but otherwise healthy and they have no contractures. 2) Most research in exercise in patients with MD or CP focuses on preventing patients from being wheelchair bound - only very little research is done in the most severely affected patients that are wheelchair bound, although many of their symptoms can potentially be ameliorated by exercise. 3) To date, research in exercise in wheelchair bound patients with MD or CP has primarily consisted of arm cycling. It has been shown to reduce BMI and improve cardiorespiratory status, endurance, muscle strength and activities of daily living, but not without complications. The upper limbs consist of small muscle groups that are easily fatigued and therefore proper cardiopulmonary fitness is difficult to obtain. The risk of upper limb overuse injuries is high, reducing patients function and activities of daily living. Presently, there is no feasible and acceptable way to exercise for this large patient group.

The investigators have tested a cycle ergometer for the lower limbs that can be used while the patients sit in their own wheelchair. It has a motor, since most patients are not able to turn the pedals themselves, and a sensor that can measure how much patients contribute to cycling. They have tested 3 wheelchair bound patients. After training, they all experienced reduced pain in lower back and glutes, less obstipation and increased energy. Surprisingly, the heart rate increased during exercise by up to 65 beats even in patients that could not turn the pedals themselves, indicating cardiovascular fitness. To test this form of exercise in a larger group of patients that are wheelchair bound due to MD or CP will be of great interest.

The aim of this project is thus:

1. to test a cycle ergometer for lower limbs in patients who are wheelchair bound due to MD or CP to find a feasible and acceptable way to exercise in order to increase health and quality of life.
2. to investigate if patients unable to move their legs will have effect of the training.

ELIGIBILITY:
Inclusion Criteria:

* Verified muscular dystrophy or cerebral palsy
* Age: Over 18 years
* Wheelchair use; can at maximum stand up for transfers and is unable to walk for more than 5 meters.

Exclusion Criteria:

* Competing disorders (as arthritis) or other muscle disorders
* Unable to use the cycle ergometer due to contractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Questionnaire on fatigue | 5 minutes
  The FSS (fatigue severity scale) will be used. Scores range from 1 to 7 with a total maximum score at 63. Lower scores mean less fatigue.
Questionnaire on pain. | 5 minutes
  A visual pain score that has been used in former studies with 3 questions with scores ranging from 1 to 10 each, 10 being the worst pain imaginable, will be used.
Questionnaire on constipation | 5 minutes
  A questionnaire made from the Danish definition of constipation will be used. Four questions will be answered "yes" or "no".
Questionnaire on quality of life, QOL | 10 minutes
  A QOL that has been used in former studies will be used. 16 questions with scores ranging from 1 (very unsatisfied) to 7 (very satisfied) will be scored.

SECONDARY OUTCOMES:
Blood sample | 5 minutes
  Change in blood sample for blood lipids, mmol/l
Blood sample | 5 minutes
  Change in blood sample for HbA1C, mmol/mol
Blood sample | 5 minutes
  Change in blood sample for Creatine kinase, U/I. This will be monitored before, in the middle and after the exercise period as a safety measure.
Ultrasound | 20 minutes
  Change in muscle cross sectional area in thigh, cm2
Ultrasound | 20 minutes
  Change in muscle fat fraction in thigh, %
Exercise test | 30 minutes
  Change in time it takes to cycle 1 km, minutes
Motorscore | 30 minutes
  Change in motor-score - MFM-32 (muscular dystrophy) or GMFM-88 (cerebral palsy)

CONTACTS AND LOCATIONS:
Overall Officials: Nanna S Poulsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen Neuromuscular Center, CNMC, depart. 8077, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carter JC, Sheehan DW, Prochoroff A, Birnkrant DJ. Muscular Dystrophies. Clin Chest Med. 2018 Jun;39(2):377-389. doi: 10.1016/j.ccm.2018.01.004. PMID 29779596
- [Background] Koman LA, Smith BP, Shilt JS. Cerebral palsy. Lancet. 2004 May 15;363(9421):1619-31. doi: 10.1016/S0140-6736(04)16207-7. PMID 15145637
- [Background] Ellapen TJ, Hammill HV, Swanepoel M, Strydom GL. The health benefits and constraints of exercise therapy for wheelchair users: A clinical commentary. Afr J Disabil. 2017 Sep 8;6:337. doi: 10.4102/ajod.v6i0.337. eCollection 2017. PMID 28936414
- [Background] Glaser RM. Arm exercise training for wheelchair users. Med Sci Sports Exerc. 1989 Oct;21(5 Suppl):S149-57. PMID 2691827
- [Background] Skalsky AJ, McDonald CM. Prevention and management of limb contractures in neuromuscular diseases. Phys Med Rehabil Clin N Am. 2012 Aug;23(3):675-87. doi: 10.1016/j.pmr.2012.06.009. PMID 22938881
- [Background] Dahlqvist JR, Poulsen NS, Ostergaard ST, Fornander F, de Stricker Borch J, Danielsen ER, Thomsen C, Vissing J. Evaluation of inflammatory lesions over 2 years in facioscapulohumeral muscular dystrophy. Neurology. 2020 Sep 1;95(9):e1211-e1221. doi: 10.1212/WNL.0000000000010155. Epub 2020 Jul 1. PMID 32611642
- [Background] Janssen TW, Beltman JM, Elich P, Koppe PA, Konijnenbelt H, de Haan A, Gerrits KH. Effects of electric stimulation-assisted cycling training in people with chronic stroke. Arch Phys Med Rehabil. 2008 Mar;89(3):463-9. doi: 10.1016/j.apmr.2007.09.028. PMID 18295624